CLINICAL TRIAL: NCT07374848
Title: An Open-label, Phase 1a/b, Multicenter Study of ZL-6201 to Evaluate Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy in Participants With Sarcoma and Selected Solid Tumors
Brief Title: Phase 1a/b Study of ZL-6201 Safety, PK, and Preliminary Efficacy in Sarcoma and Selected Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Collaborators: Zai Lab (US) LLC (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZL-6201-001
Record Dates: First submitted 2025-12-15; First posted 2026-01-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors; Sarcomas
Keywords: Sarcoma; Solid Tumors; Phase1; Antibody-Drug Conjugate (ADC); Leucine-Rich Repeat-Containing protein 15 (LRRC15)
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZL-6201 (Experimental): ZL-6201 as a single agent
  Interventions: Drug: ZL-6201

INTERVENTIONS:
Drug: ZL-6201 — ZL-6201 as a single-agent

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of investigational study drug ZL-6201 for treating sarcoma and solid tumors cancer.

DETAILED DESCRIPTION:
An Open-label, Phase 1a/b, Multicenter Study of ZL-6201 to Evaluate Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy in Participants with Sarcoma and Selected Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women ≥18 years of age at the time of signing the ICF with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and a life expectancy > 3 months
* Participants must have histologically confirmed and documented diagnosis of locally advanced unresectable and/or metastatic sarcoma or a selected solid tumor
* Participants must be willing to undergo a tumor biopsy prior to start of treatment or provide archived tumor tissue sample
* Participants with sarcoma should have received no more than 2 lines of previous systemic therapies in the metastatic setting
* Participants with selected epithelial solid tumors should have received no more than 3 lines of previous systemic therapy in the metastatic/relapsed refractory setting
* Participants must have at least one measurable target lesion as defined by RECIST v1.1
* Adequate organ and marrow function as listed per protocol
* Must be negative for HIV, HBV, and HCV

Exclusion Criteria:

* Participants with another known malignancy that has required treatment within the last 2 years
* Symptomatic central nervous system (CNS) metastasis, and/or those requiring therapy with corticosteroids or anticonvulsants to control associated symptoms
* Participants with leptomeningeal metastasis
* Most recent systemic anti-cancer treatment or investigational products/devices less than 3 weeks
* Prior treatment with a topoisomerase-1 inhibitor antibody drug conjugate
* Impaired cardiac function or clinically significant cardiac disease within the last 3 months before administration of the first dose of the study treatment
* Clinically significant pulmonary disease including autoimmune, connective tissue, or inflammatory conditions
* Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities | 1 cycle of study treatment (each cycle is 21 days)
  Number of subjects with dose limiting toxicities (DLTs) through dose escalation only.
Incidence of Treatment Emergent Adverse Events | 36 months
  Number of subjects with treatment-emergent adverse effects through dose escalation and expansion.
Incidence of Serious adverse events | 36 months
  Number of subjects with Serious Adverse Events through dose escalation and expansion.
Number of participants with clinical laboratory abnormalities | 36 months
Number of participants with vital sign abnormalities | 36 months
  Vitals will be measured in Riva Rocci (RR) in mmHG and Pulse in beats per minute
Number of participants with electrocardiogram (ECG) abnormalities | 36 months
  ECG will be measured in ECG intervals (QT and QTc with Fridericia correction, and PR), QRS duration, and heart rate will be tested and analyzed.

SECONDARY OUTCOMES:
ORR per RECIST 1.1 | 36 months
  Objective Response Rate (ORR) is defined as the proportion of participants who have a best response of confirmed partial response (PR) or confirmed complete response (CR) to study treatment per RECIST v1.1 by investigator assessment through dose escalation and expansion.
Duration of Response per RECIST 1.1 | 36 months
  Duration of Response is defined as the time from the first assessment of CR or PR to the first assessment of progression disease (PD) by investigator per RECIST 1.1 or death due to any cause (whichever occurs first) through dose escalation and expansion.
PFS per RECIST 1.1 | 36 months
  Progression-Free Survival (PFS) is defined as the time from first dosing date to the first documented PD by investigator per RECIST 1.1 or death for any reasons (whichever occurs first) through dose escalation and expansion.
DCR per RECIST 1.1 | 36 months
  Disease Control Rate (DCR) is defined as the proportion of participants who have a best response of confirmed CR, confirmed PR, or SD per RECIST 1.1 by investigator assessment through dose escalation and expansion.
PK characteristics of ZL-6201 (ADC conjugate), total antibody | 36 months
  Pharmacokinetics: Total Antibody of ZL-6201
PK characteristics of ZL-6201 (ADC conjugate), unconjugated payloads | 36 month
  Pharmacokinetics: Unconjugated payloads of ZL-6201

CONTACTS AND LOCATIONS:
Locations (1):
- Zai Lab Site 02006, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No